CLINICAL TRIAL: NCT06255769
Title: Identification of Myocardial Ischemia With Magnetocardiography Using Single Photon Emission Computed Tomography (SPECT) as a Reference Standard
Brief Title: Diagnosis of Myocardial Ischemia With MCG Using SPECT as a Reference Standard
Status: Recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Chongqing Emergency Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MCG-SPECT
Record Dates: First submitted 2024-01-30; First posted 2024-02-13 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Chest Pain; Stenosis; Myocardial Ischemia
MeSH Terms: conditions — Chest Pain; Constriction, Pathologic; Myocardial Ischemia | interventions — Magnetocardiography; Tomography, Emission-Computed, Single-Photon

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Magnetocardiography — Magnetocardiography
Device: Single photon emission computed tomography (SPECT) — Single photon emission computed tomography (SPECT)

SUMMARY:
This is a prospective clinical study aiming to investigate the efficacy of Magnetocardiography (MCG) in detecting myocardial ischemia in patients of a suspected non-ST-elevation-acute coronary syndrome (NSTE-ACS) by using Single photon emission computed tomography (SPECT) as the gold standard for determining the presence and severity of myocardial ischemia.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older;
* Patients with symptoms of myocardial ischemia such as angina pectoris, who have CAG showing <70% stenosis at the most severe site or CTA showing non-severe stenosis
* Signed informed consent.

Exclusion Criteria:

* Patients with absolute or relative contraindications to SPECT-loaded myocardial perfusion, including acute myocardial infarction within 48 hours, significant left main coronary artery stenosis, bronchial asthma, and adenosine injection allergy;
* Patients with Non-ischemic dilated cardiomyopathy, or hypertrophic cardiomyopathy, or moderate or severe valvular disease;
* Patients with Hemodynamic instability (systolic blood pressure<90 mmHg, or who requires vasoactive drugs), or patients with tachyarrhythmia, Ⅱdegree atrioventricular block and above that have not returned to normal;
* Patients who have severe renal abnormality with eGFR <30 ml/min, or patients who are on dialysis;
* Patients with malignant tumors with predicted survival of less than 1 year;
* Pregnant or breastfeeding women;
* Patients who are unable to enter the MCG device, who are unable to perform MCG examination due to interference from metal implants or other reasons, or who are deemed by the investigators to be unsuitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chest pain patients who have CAG showing <70% stenosis at the most severe site or CTA showing non-severe stenosis
Sampling Method: Non-Probability Sample
Enrollment: 228 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of MCG to detect myocardial ischemia using SPECT as a reference standard. | from the date of enrollment until the date of discharge, up to 30 days
  Sensitivity, specificity, and area under the ROC curve are performed for assessing the efficacy.

SECONDARY OUTCOMES:
Efficacy of MCG to detect myocardial ischemia in patients with coronary stenosis <50% (Ischemia with no obstructive coronary artery, INOCA) | from the date of enrollment until the date of discharge, up to 30 days
  Sensitivity, specificity, and area under the ROC curve are performed for assessing the efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Yuguo Chen, Professor, Principal Investigator — Qliu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China